CLINICAL TRIAL: NCT01169844
Title: An Open Label Non-randomized Extension Study to Evaluate the Safety and Tolerability of AIN457 (Anti Interleukin-17 Monoclonal Antibody) in Patients With Psoriatic Arthritis
Brief Title: Safety and Tolerability of AIN457 in Adults (18-65 Years) With Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A2206E1
Record Dates: First submitted 2010-07-14; First posted 2010-07-26 (Estimated); Results first posted 2021-05-27 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; IgG1K monoclonal antibody; Interleukin -17A neutralizing
MeSH Terms: conditions — Arthritis, Psoriatic

ARMS (2):
- AIN457/AIN457 3 mg/kg. (Experimental): Participants who were treated with secukinumab 2x10 mg/kg during the core study were treated with secukinumab at 3mg/kg infused intravenously every 4 weeks during the extension study, over a total period of 52 weeks.
  Interventions: Biological: AIN457A
- Placebo/AIN457 3 mg/kg. (Placebo Comparator): Participants who were treated with placebo during the core study were treated with secukinumab at 3mg/kg infused intravenously every 4 weeks during the extension study, over a total period of 52 weeks.
  Interventions: Biological: AIN457A; Other: Other

INTERVENTIONS:
Biological: AIN457A
Other: Other
  Arms: Placebo/AIN457 3 mg/kg.

SUMMARY:
This study is designed as an extension study to the proof-of-concept trial CAIN457A2206 in patients with psoriatic arthritis and aims to provide continuous treatment with AIN457 for patients in the core trial, to obtain safety and tolerability information. The study will address the evaluation of efficacy following doses of 3 mg/kg AIN457 given every 4 weeks over a period initially up to 6 months (Part 1) and based on the risk/benefit balance of AIN457 in psoriatic arthritis a decision will be made as to whether or not to continue dosing for another 6 month period (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated and completed the core CAIN457A2206 study up to and including the end of the study (EoS) Visit, i.e. Visit 16 (Week 24), were allowed to enter the extension study upon signing informed consent.
* Patients who discontinued the core study due to unsatisfactory therapeutic effect at their Visit 14 (Week 16) or a later visit could enter the extension study within three weeks of completing the study discontinuation visit of the core study, provided that at their discontinuation visit they met the criteria below. Patients who did not enter the extension study within 3 weeks of completing the study discontinuation visit of the core study, were to have an additional baseline visit (Visit 17) and required to meet the criteria below:
* The number of tender joints was the same or more than the core study baseline; or,
* The number of swollen joints was the same or more than the core study baseline; or,
* There was no improvement compared with the core study baseline in at least three of the following five domains: patient global assessment, physician global assessment, patient pain assessment, Health Assessment Questionnaire and CRP

Exclusion Criteria:

* Patients for whom continued treatment with AIN457 is not considered appropriate by the treating physician.
* Patients who were non-compliant or who demonstrated a major protocol deviation in the core CAIN457A2206 study.
* Patients who discontinued from the core CAIN457A2206 study before Visit 14 (Week 16), and patients who completed the core study or discontinued the core study more than 2 weeks before the baseline visit.
* Pregnant or lactating women
* Presence of active infection
* Positive PPD or HIV test in patients where repeated testing was deemed appropriate due to their risk profile

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Hamburg, Germany
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam, DE
  - Novartis Investigative Site, Meerssen, KR
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 42 patients were randomized in the (CAIN457A2206) core study, of which 28 patients enrolled into the (CAIN457A2206E1) extension study.
Period: Overall Study
Arm/Group | AIN457/AIN457 3 mg/kg. | Placebo/AIN457 3 mg/kg
Started | 19 | 9
Completed | 14 | 8
Not Completed | 5 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Patient withdrew consent | 4 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457/AIN457 3 mg/kg | Placebo/AIN457 3 mg/kg | Total
Number analyzed (Participants) | 19 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (10.96) | 47.9 (6.81) | 46.3 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Predominant race: Caucasian | 19 | 8 | 27
  Predominant race: Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Other | 19 | 8 | 27
  Ethnicity: Hispanic/Latino | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: Up to 64 weeks (End of the Study Treatment)
Population: The safety population consisted of all randomized patients who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457/AIN457 3 mg/kg | Placebo/AIN457 3 mg/kg
Number analyzed (Participants) | 19 | 9
Participants
  Serious Adverse Events | 5 | 2
  Death | 0 | 0

2. Secondary Outcome: Total IL-17 Concentration in Blood at Steady-state
Description: Total IL-17 concentration was not reported due to assay limitations.
Time Frame: Up to 64 weeks
Population: No participants were evaluated as IL-17 concentration was not reported due to assay limitations
Arm/Group | AIN457/AIN457 3 mg/kg | Placebo/AIN457 3 mg/kg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Serum Concentration Measured at Steady State
Description: This outcome measure is assessing AIN457 Mean Serum Concentration Measured at Steady State. A competitive ELISA method was used for bioanalytical analyses and the anticipated LLOQ is 80 nanograms/mL serum.
Time Frame: Weeks 0, 8, 16, 20, 24, 28, 32, 36, 40 and at 4 and 12 weeks after the last administration at Week 52.
Population: All participants from the safety set with quantifiable pharmacokinetic (PK) measurements and no major protocol deviations with impact on PK data were included in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: Microgram/millilitre (μg/mL)
Arm/Group | AIN457/AIN457 3 mg/kg | Placebo/AIN457 3 mg/kg
Number analyzed (Participants) | 19 | 9
Microgram/millilitre (μg/mL)
  0/pre-inf: number analyzed (Participants) | 14 | 9
  0/pre-inf | 2.76 (4.73) | 0.00 (0.00)
  0/post-inf: number analyzed (Participants) | 15 | 9
  0/post-inf | 80.0 (17.7) | 68.8 (19.1)
  8/pre-inf: number analyzed (Participants) | 12 | 7
  8/pre-inf | 29.6 (10.3) | 19.5 (7.68)
  8 /post-inf: number analyzed (Participants) | 12 | 7
  8 /post-inf | 99.7 (22.1) | 88.9 (25.5)
  16/pre-inf: number analyzed (Participants) | 9 | 8
  16/pre-inf | 32.9 (12.1) | 23.3 (10.3)
  16/post-inf: number analyzed (Participants) | 9 | 8
  16/post-inf | 110 (25.3) | 82.9 (24.7)
  20/pre-inf: number analyzed (Participants) | 12 | 8
  20/pre-inf | 31.3 (9.00) | 25.4 (13.0)
  20/post-inf: number analyzed (Participants) | 10 | 8
  20/post-inf | 111 (29.9) | 85.5 (19.9)
  24/pre-inf: number analyzed (Participants) | 11 | 8
  24/pre-inf | 37.2 (11.9) | 25.5 (11.6)
  24/post-inf: number analyzed (Participants) | 11 | 8
  24/post-inf | 109 (24.5) | 89.1 (23.2)
  28/pre-inf: number analyzed (Participants) | 8 | 7
  28/pre-inf | 37.4 (10.2) | 22.1 (9.45)
  28/post-inf: number analyzed (Participants) | 8 | 6
  28/post-inf | 122 (20.2) | 96.9 (18.5)
  32/pre-inf: number analyzed (Participants) | 9 | 7
  32/pre-inf | 37.4 (13.0) | 26.7 (8.05)
  32/post-inf: number analyzed (Participants) | 8 | 7
  32/post-inf | 112 (15.1) | 92.8 (23.2)
  36/pre-inf: number analyzed (Participants) | 10 | 6
  36/pre-inf | 33.4 (9.49) | 27.3 (7.06)
  36/post-inf: number analyzed (Participants) | 9 | 7
  36/post-inf | 109 (24.4) | 88.9 (13.9)
  40/pre-inf: number analyzed (Participants) | 10 | 8
  40/pre-inf | 46.4 (28.2) | 28.7 (9.00)
  40/post-inf: number analyzed (Participants) | 10 | 7
  40/post-inf | 84.8 (30.5) | 105 (24.9)
  56: number analyzed (Participants) | 12 | 8
  56 | 33.8 (8.93) | 31.6 (7.62)
  64: number analyzed (Participants) | 10 | 5
  64 | 11.0 (3.46) | 10.3 (8.31)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment (Week 52), and continued up to Week 64
Arm/Group | AIN457/AIN457 3 mg/kg | Placebo/AIN457 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/19 | 2/9
Other Adverse Events (participants affected / at risk) | 19/19 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457/AIN457 3 mg/kg (N=19) | Placebo/AIN457 3 mg/kg (N=9)
Myocardial infarction (Cardiac disorders) | 0 | 1
Viral sinusitis (Infections and infestations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Sciatica (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457/AIN457 3 mg/kg (N=19) | Placebo/AIN457 3 mg/kg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 3
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 4
Onychomycosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Blood immunoglobulin G increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 2
Weight decreased (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.